CLINICAL TRIAL: NCT06275672
Title: TREAT INTERACT: Implementing a User Involved Education- and Health System Interactive Task-shifting Approach for Child Mental Health Promotion in Uganda
Brief Title: Implementing an Education- and Health System Task-shifting Approach for Child Mental Health Promotion in Uganda
Acronym: TREAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Makerere University (Other); University of Bergen (Other); Norwegian Institute of Public Health (Other Government); Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: TREAT INTERACT
Record Dates: First submitted 2023-12-28; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue; Stigma, Social; Child Development; Child Abuse
Keywords: Adolescent; Child; Global mental health; Implementation; Low- and middle income countries; Primary schools; Task shifting; Teachers; Uganda
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial to randomize 18 schools into six cohorts of three schools incrementally.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Active Comparator): An Ugandan adapted version of the mhGAP-IG child and adolescent mental health module will be used for identification, assessment, and management of common mental disorders in children and adolescents at primary schools.
  Interventions: Other: Adapted version of the mhGAP-IG
- Cohort 2 (Active Comparator): Same as arm 1
  Interventions: Other: Adapted version of the mhGAP-IG
- Cohort 3 (Active Comparator): Same as arms 1-2
  Interventions: Other: Adapted version of the mhGAP-IG
- Cohort 4 (Active Comparator): Same as arms 1-3
  Interventions: Other: Adapted version of the mhGAP-IG
- Cohort 5 (Active Comparator): Same as arms 1-4
  Interventions: Other: Adapted version of the mhGAP-IG
- Cohort 6 (Active Comparator): Same as arms 1-5
  Interventions: Other: Adapted version of the mhGAP-IG

INTERVENTIONS:
Other: Adapted version of the mhGAP-IG — An Ugandan adapted version of the mhGAP-IG CAMH module for identification, assessment, and management of common mental disorders in children and adolescents. The mhGAP-IG CAMH module further details six different protocols for the management of these mental health problems, primarily based on psychosocial and systemic interventions. The described psychosocial interventions can also be provided as general prevention for children with subclinical problems. Lastly, the module guides further follow-up assessment. Experts identified by the Ministry of Health will train trainers who train and follow-up teachers and health personnel receiving the intervention.

SUMMARY:
This study will adapt a school version (mhGAP-IGs) of the World Health Organization´s (WHO) "Mental Health Gap Action Programme Intervention Guide" (mhGAP). Both teachers and health workers will receive training in mhGAP, and systems for collaboration between the school and health sector as well as other relevant stakeholders will be developed and integrated. The project is conducted in close collaboration with key stakeholders from the Ministry, the health and education sector, the police, and religious leaders. The aim is to increase mental health literacy among school staff, facilitate a healthy school environment, and increase detection of mental health needs among primary school aged children.

DETAILED DESCRIPTION:
Background: Mental and neuropsychological disorders make up approximately 14 percent of the total health burden globally, with 80% of the affected living in low- and middle-income countries (LMICs). In these countries, more than 90% of children cannot access mental health services, therefore service strengthening is warranted. The main objective of the TREAT INTERACT study is to adapt, implement and evaluate the impact of a novel, intersectoral treatment interactive approach to prevent, identify, refer, and treat mental health problems in children and adolescents through a user centered task-shifting adaptation and implementation of the World Health Organization (WHO) Mental Health Gap Action Programme (mhGAP) Intervention Guide (mhGAP-IG) for primary school staff in Mbale, Eastern Uganda. In this study the aims are to: 1) Adapt the mhGAP-IG to primary school settings, 2) Implement the adapted module-based school program and investigate effective implementation strategies and teacher, student, and caregiver outcomes, 3) Develop, implement and evaluate an intersectoral supervision, referral and communication model between the health and education sectors, and 4) Develop sustainable and scalable implementation advice and guidelines with policymakers.

Methods: This project is a pragmatic mixed-methods hybrid Type II Implementation-Effectiveness study utilizing a co-design approach. The main study will utilize a stepped-wedged design with phased implementation where participating schools will be randomized to intervention initiation. Those not yet randomized to the intervention will serve as "controls". There will be six starting sequences and three schools will be randomized to intervention initiation at each randomization interval. In addition, other quantitative designs including a nested prospective cohort, case control studies, cross-sectional studies in addition to qualitative research will strengthen the necessary components for successful implementation and evaluation.

Population: Teachers are the primary participants in the trial. In addition, data will be collected from health personnel, school leadership, pupils and their caregivers.

Outcomes: Implementation outcomes include detection, reach, sustainability and service delivery to children and adolescents in need of the mhGAP from the school and health sectors. Main client outcomes include teachers´ mental health literacy, stigma and violence towards the school children. Child and caregiver outcomes will include mental health status, mental health literacy, and help-seeking behavior.

Discussion: This study will provide knowledge on implementation and sustainability of mental health programs relevant for children in primary schools in line with current WHO guidelines.

ELIGIBILITY:
Inclusion Criteria:

* A teacher/ staff member at a preselected TREAT INTERACT primary school in Mbale.
* Child-caregiver pairs are eligible when a learner is enrolled in a selected primary school in Mbale, the child has a caregiver living with him or her and provides ascent, and the caregiver with a child in the selected school providing informed consent.

Exclusion Criteria:

* Not part of preselected primary school
* Lack of informed consent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reach questionnaire, developed by the project group | Through study completion, an average of 1.5 years
  For teachers. Proportion of children reached by the program. Consist of one question: "Have you ever referred a child at school to the health system?" If no (scored 0), no further questions are asked. If yes (scored 1), an additional 5 questions follows (e.g., "If yes, have any of these referrals to the health system been because of a mental health problem?")
The Program Sustainability tool (Finch et al., 2013) | Through study completion, an average of 1.5 years
  For teachers. 22 items measuring the following:
  * Financial stability
  * Organizational Support
  * Staff Retention:
  * Program Integration
  * Stakeholder Perceptions
  * Program Outcomes and Impact
  It is scored from 0 (little to no extent) to 7 (to a very great extent). A summed score is created (a minimum score of 0 and a maximum score of 154, where a higher score mean a better outcome)
Service measure on access to mental health care, developed by the project group | Through study completion, an average of 1.5 years
  For teachers. 21 items measuring the following dimention of Service Utilization will be created during the mapping process:
  * Wait Times
  * Geographical Accessibility
  * Affordability
  * Equity and Disparities
  * Satisfaction and Perceived Access
  * Referral Patterns
  * Availability of Services Scored 0 (never) to 4 (at least once a year). A summed score is created (a minimum score of 0 and a maximum score of 105, where a higher score mean a better outcome)
Attitudes about Child Mental Health (Perceived Discrimination-Devaluation (Link et al., 1987) questionnaire | Through study completion, an average of 1.5 years
  For teachers. 10 items measuring stigma and mental health literacy.
  Scored from 1 (strongly disagree) to 7 (strongly agree). A summed score is created (a minimum score of 0 and a maximum score of 70, where a higher score mean a better outcome)
The dimensions of discipline inventory, school (DDI; Strauss & Faucher, 2007) | Through study completion, an average of 1.5 years
  For children. 11 items measuring incidents of teacher violence. Scored from 0 (never) to 4 (at least once a year). A summed score is created (a minimum score of 0 and a maximum score of 44, where a higher score mean a worse outcome)
Treatment at home, developed by the project group, by inspiration from our siste project "TREAT C-AUD") | Through study completion, an average of 1.5 years
  For children. 10 items measuring treatment at home. Scoring instructions will be deveoped during the mapping process.

SECONDARY OUTCOMES:
The Implementation Quality Questionnaire (Bogen, 2020) | Through study completion, an average of 1.5 years
  For teachers and school staff. 26 questions on the perception of acceptability, appropriateness, feasibility, ownership, school climate and user participation. Scored from 1 (strongly disagree) to 7 (strongtly agree). A summed score is created, as well as a score for each dimention (a minimum score of 0 and a maximum score of 182, where a higher score mean a better outcome)
Fidelity Scale, developed by the project group | Through study completion, an average of 1.5 years
  For teachers. A scale to measure the fidelity to the intervention, including adaptations and modifications will be developed as part of the mapping process.
General Health Questionnaire (GHQ; Goldberg, 1970) | Through study completion, an average of 1.5 years
  For teachers. 12 items measuring personal mental health, scored 1 (better than usual) to 4 (much less than usual). A summed score is created (a minimum score of 0 and a maximum score of 48, where a higher score mean a worse outcome)
Attitudes on Gender Norms (Waszak et al., 2000) questionnaire | Through study completion, an average of 1.5 years
  For teachers and caregivers. 10 items measuring tteacher reported gender norms. Scored 0 (disagree) or 1 (agree). A summed score is created (a minimum score of 0 and a maximum score of 10, where a higher score mean a better outcome)
Help-seeking behaviour, developed by the project group after inspiration from Yifeng et al., 2022 | Through study completion, an average of 1.5 years
  For caregivers. Help seeking behaviour is measured by the following question: At any point during the past 3 months, did you ever speak to a health professional about any mental health problem or concern? Scored from 1 ( did not have any mental health problem or concern) to 4 (I decided not to speak to a health professional although I am concerned about my mental health).
Pediatric Symptom Checklist (PSC-17; Jellinek et al., 1998) | Through study completion, an average of 1.5 years
  For children. 17 items measuring child mental health. Scored 0 (never) to 2 (often). A summed score is created(a minimum score of 0 and a maximum score of 34, where a higher score mean a worse outcome)
Teacher Support Scale (TSS; Metheny, McWhirter, & O'Neil, 2008) | Through study completion, an average of 1.5 years
  For children. 21 items measuring child-reported support from teachers. Scored from 1 (disagree) to 3 (agree). A summed score is created (a minimum score of 21 and a maximum score of 63, where a higher score mean a better outcome)
Teacher violence scale (Piskin et al, 2014) | Through study completion, an average of 1.5 years
  For children. 29 items on teacher violence. Scored from 0 (never) to 5 (every day) (a minimum score of 0 and a maximum score of 145, where a higher score mean a worse outcome)
The dimensions of discipline inventory, home (DDI; Strauss & Faucher, 2007) | Through study completion, an average of 1.5 years
  For children. 7 items measuring discipline at home. Scored from 0 (never) to 4 (at least once a year) (a minimum score of 0 and a maximum score of 28, where a higher score mean a worse outcome)
The Implementation Leadership Scale (Aarons, Ehrhart, et al., 2014) | Through study completion, an average of 1.5 years
  For teachers. 12 items measuring the following subscales: Proactive, knowledgeable, supportive, perservant, and available. Scored 0 (not at al) to 4 (to a very great extent). A summed score is created (a minimum score of 0 and a maximum score of 48, where a higher score mean a better outcome)
Organizational Readiness for Implementing Change (Shea et al., 2014) | Through study completion, an average of 1.5 years
  For teachers and scool staff. 12 items measuring change efficacy. Scored from 1 (strongly disagree) to 5 (strongly agree). A summed score is created (a minimum score of 12 and a maximum score of 60, where a higher score mean a better outcome)
Teacher concerns about child mental health, developed by the project group, after inspiration from Yifeng et al., 2022 | Through study completion, an average of 1.5 years
  For teachers. 7 items measuring concerns, referrals, and support. Each question is scored individually (both yes/no, number response, and qualitative resonse)
Provider Report of Sustainment Scale (PRESS) (Moullin et al., 2021) (PRESS): development and validation (PRESS; Moullin et al., 2021) | Through study completion, an average of 1.5 years
  For teachers. 3 items measuring if staff use the intervention. Scored from 0 (not al all) to 4 (to a very great extent). A summed score is created (a minimum score of 0 and a maximum score of 12, where a higher score mean a better outcome)
Mental health knowledge (Evans-Lacko et al., | Through study completion, an average of 1.5 years
  For caregivers. 17 items measuring caregiver mental health literacy. Scored from 1 (disagree strongly) to 6 (agree strongly). A summed score is created (a minimum score of 17 and a maximum score of 102, where a higher score mean a better outcome)
AUDIT scale (WHO) | Through study completion, an average of 1.5 years
  For caregivers. 11 items measuring alcohol use by caregivers. Scoring will be decided in accordance to the RQ later in the mapping process.
Child alcohol use, developed by the project group | Through study completion, an average of 1.5 years
  For children. 5 items measuring child alcohol use (e.g., Have you ever had a drink of alcohol rather than a few sips?). Scored individually (numeric or yes/no).
Child mental health - Pediatric symptoms (Jelinek et al.) | Through study completion, an average of 1.5 years
  For children. 17 self-report questions on child mental health. Scored from 0 (never) to 2 (often). A summed score is created (a minimum score of 0 and a maximum score of 34, where a higher score mean a worse outcome)
Perceived teacher support and its influence on adolescent career development (Metheny et al., 2008) | Through study completion, an average of 1.5 years
  For children. 21 items scored from 1 (disagree) to 3 (agree). A summed score is created (a minimum score of 21 and a maximum score of 63, where a higher score mean a better outcome)
Sexual violence, developed by the project group | Through study completion, an average of 1.5 years
  For children. 9 items on experiences of sexual violece. Scored from 0 (no) to 3 (every term). A summed score is created (a minimum score of 0 and a maximum score of 27, where a higher score mean a worse outcome)
Dimensions of discipline inventory (DDI; Straus and Fauchier, 2007) | Through study completion, an average of 1.5 years
  For children. 7 items measuring corporal punishment. Scored from 0 (never) to 4 (at least once a year). A summed score is calculated (a minimum score of 0 and a maximum score of 28, where a higher score mean a worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ane-Marthe Solheim Skar, Principal Investigator — Norwegian Center for Voilence and Traumatic Stress Studies
Locations (1):
- Nowegian Center for Violence and Traumatic Stress Studies, Oslo, Norway

REFERENCES:
- [Derived] Skar AS, Engebretsen IMS, Braathu N, Aber H, Baekkelund H, Kuhl MJ, Mukisa M, Nalugya JS, Skokauskas N, Skylstad V, Wentzel-Larsen T; TREAT research consortium; Babirye JN. Study protocol for a stepped-wedge implementation study investigating the intersectoral collaboration of implementering the TREAT INTERACT intervention for primary school teachers and the mhGAP for health care workers for child mental health promotion in Uganda. Trials. 2024 Jul 9;25(1):465. doi: 10.1186/s13063-024-08312-5. PMID 38982328